CLINICAL TRIAL: NCT05827601
Title: Active Surveillance of Influenza Virus Zoonotic Transmission Events: a Pilot Study in Belgium
Brief Title: Zoonotic Influenza Surveillance in Belgium
Acronym: ZOOIS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Cyril Barbezange (Other Government)
Collaborators: Sciensano (Other Government); Belgian Federal Public Service, Food Chain Safety and Environment (Other Government); Agentschap Zorg en Gezondheid (Unknown)
Responsible Party: Sponsor-Investigator, Cyril Barbezange, Head of Belgian National Influenza Centre, Sciensano
Organization: Sciensano (Other Government)
Other Study IDs: ZOOIS-23-24
Record Dates: First submitted 2023-03-30; First posted 2023-04-25 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — Respiratory Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — respiratory specimens will be registered and stored in the Biobank for 10 years after the end of the study, and could be tested for other pathogens but they will not be used for human genetic or biomarker analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Avian Influenza Outbreak Farms: People involved in outbreak management, ranging from poultry farm owners and their family to inspectors through veterinarians and cullers/cleaners, will be invited to take part in the study at the earliest step possible after outbreak detection. Self sampling by nasopharyngeal swab will be requested every 2 days during 2 weeks.
  Interventions: Diagnostic Test: respiratory specimen; Diagnostic Test: serum
- Poultry Farm Sentinel Network: People working in poultry farms and in contact with animals will be invited to join the cohort. Self sampling by nasopharyngeal swab will be requested every 2 weeks for the whole duration of the study.
  anticipated: 15
  Interventions: Diagnostic Test: respiratory specimen
- Wild bird/life Rehabilitation Centre Sentinel Network: People working in wild bird/life rehabilitation centers and in contact with animals will be invited to join the cohort. Self sampling by nasopharyngeal swab will be requested every 2 weeks for the whole duration of the study.
  anticipated: 25
  Interventions: Diagnostic Test: respiratory specimen
- Pig Industry Veterinarian Sentinel Network: Veterinarians working in the pig industry and in contact with animals will be invited to join the cohort. Self sampling by nasopharyngeal swab will be requested every 2 weeks for the whole duration of the study.
  anticipated: 15
  Interventions: Diagnostic Test: respiratory specimen

INTERVENTIONS:
Diagnostic Test: respiratory specimen — participants will perform self-sampling with a nasopharyngeal swab
Diagnostic Test: serum — participants will be invited to get a blood sample taken by a general practitioner or to perform a self sampling of capillary blood
  Groups: Avian Influenza Outbreak Farms

SUMMARY:
The project aims at implementing a more pro-active surveillance of potential transmission of influenza viruses to humans (zoonotic transmission). Clinical surveillance of influenza in humans and avian species is well organized and has been operating for decades, but currently there is no pro-active systematic surveillance of potential transmission of animal (avian or swine) influenza viruses to humans, only follow-up of people showing clinical symptoms. People working with potentially infected animals have the highest risk. Moreover, they can represent the first steps in a pandemic: if the virus adapts to humans, infected workers could potentially spread the virus to other people.

Currently, highly pathogenic clade2.3.4.4b H5 avian influenza viruses are continuously circulating in wild birds in Belgium and the number of introduction in poultry farms has raised, increasing the contact opportunities with high viral concentrations. Several reports of suspected human infection have been made by different countries. In addition, the virus was detected in sick non-human mammals. The large circulation in wild birds thus represents an increase risk of spill-over to mammalian species, including humans, (by contact directly with wild birds, or via outbreaks in poultry). This increased opportunity for accidental spillover to new host species increases the chances for the avian virus to adapt to mammals, including humans.

Likewise, there have also been an increased number of human cases of swine influenza reported by several European countries. A pro-active surveillance aiming at also detecting asymptomatic infections would allow an early detection of transmission that could help to prevent a new pandemic.

As a piloting approach during this specific project, some dedicated sentinel networks among at-risk workers will be initiated: people in poultry farms involved with the management of outbreaks of highly pathogenic avian influenza; people working at bird (or more generally wild life) rehabilitation centres or poultry farms; veterinarians working in pig farms/slaughterhouses.

ELIGIBILITY:
Inclusion Criteria:

* worker or volunteer of one of the targeted groups at one of the selected sites and accepting to take part in the study
* to have regular contacts with animals within job/activity framework
* being committed to take the regular samples

Exclusion Criteria:

- people who had a broken nose might have difficulties to perform self-swabbing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Workers or volunteers of one of the targeted groups within the sites that accept to take part in the study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of sentinel participants positive for a non-seasonal influenza virus | every 2 weeks through study completion (December 2024)
  result of RT-qPCR test to detect and characterize non-influenza viruses
Number of outbreak participants positive for a non-seasonal influenza virus | every 2 days during 2 weeks after enrollment
  result of RT-qPCR test to detect and characterize non-influenza viruses

SECONDARY OUTCOMES:
Number of outbreak participants with seroconversion against a non-seasonal influenza virus | at enrollment and about 4 weeks after
  result of inhibition of haemagglutination or seroneutralisation assay

CONTACTS AND LOCATIONS:
Locations (1):
- Sciensano, Brussels, Belgium